CLINICAL TRIAL: NCT07234591
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of a TYK2 Inhibitor in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate Effectiveness and Safety of a TYK2 Inhibitor in Subjects With Moderate to Severe Plaque Psoriasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Usynova Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN101
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Plaque Psoriasis; Moderate to Severe Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- dose level 1 (Experimental)
  Interventions: Drug: Tyk2 inhibitor
- dose level 2 (Experimental)
  Interventions: Drug: Tyk2 inhibitor
- dose level 3 (Experimental)
  Interventions: Drug: Tyk2 inhibitor
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tyk2 inhibitor — Specific dose of Tyk2 inhibitor on specific days
  Arms: dose level 1; dose level 2; dose level 3
Drug: Placebo — Specified dose of Placebo on specified days.
  Arms: placebo

SUMMARY:
A Study to evaluate efficacy and safety in subjects with moderate to severe Plaque Psoriasis treated with a TYK2 Inhibitor for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Male and female, ages 18 to 70 years
* Body weight >40 kg, body mass index (BMI) of 18 to 40 kg/m2
* Clinical diagnosis of plaque psoriasis for ≥6 months before the Baseline visit
* Women of childbearing potential (WOCBP) and males who are sexucally active must agree to follow instructions for method(s) of contraception.

Exclusion Criteria:

* Diagnosed with non-plaque psoriasis
* Previously received tyrosine kinase 2 (TYK2) inhibitors
* Previously received other psoriasis treatments such as biological agents, immunoregulators, or hormonal drugs within a specific period before administration, and the investigator deems it may affect the immunity of the subjects
* Has participated in any clinical trials within 30 days or 5 half-lives of the drug before the first administration, or currently undergoing visits for other clinical trials;
* Has history of chronic disease that may affect the study, or acute or chronic severe infectious diseases, such as a history of active or inadequately treated latent tuberculosis infection, severe bone or joint infections within 6 months before screening, and other acute infectious diseases.
* Has known or suspected skin or systemic autoimmune diseases other than psoriasis and psoriatic arthritis;
* Other conditions that the investigator deems unsuitable for participation in this study.

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
The Percentage of Participants Experiencing a 75% Improvement (Reduction From Baseline) in PASI Score (PASI-75 Response Rate) on Week 12 | Baseline to Week 12

SECONDARY OUTCOMES:
Percentage of Participants With PASI-90, PASI-100 on Week 12 | Baseline to Week 12
Percentage of Participants on Week 12 With sPGA Score of 0 or 1 (sPGA0/1 Response Rate) | Baseline to Week 12
Change From Baseline in DLQI Scores to Week 12 | Baseline to Week 12
Change From Baseline in BSA to Week 12 | Baseline to Week 12
Number of Participants With Adverse Events | From enrollment to Day 112
Mean steady-state plasma concentration of the drug (Cav,ss) | Day 1, Day 8, Day 15, Day 29, Day 57, Day 84
Steady-state trough plasma concentration of the drug (Ctrough, ss) | Day 1, Day 8, Day 15, Day 29, Day 57, Day 84
The area under the steady-state blood drug concentration-time curve (AUCss) | Day 1, Day 8, Day 15, Day 29, Day 57, Day 84

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Skin Disease Hospital, Shanghai, China